CLINICAL TRIAL: NCT01386190
Title: Impact of Exercise on Body Composition in Premature Infants: New Approaches
Brief Title: Impact of Exercise on Body Composition in Premature Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Non applicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01H110163-01A1 [2011-8156]; HS # 2011-8156 (Other: IRB #)
Record Dates: First submitted 2011-06-21; First posted 2011-06-30 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Body Composition, Beneficial
Keywords: preterm infant, body composition, exercise
MeSH Terms: conditions — Glucocorticoid Receptor Deficiency; Premature Birth; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Group (Experimental): Caregivers will be taught progressive exercises to use with their infants from hospital discharge to 1 year of age.
  Interventions: Other: Exercise/Social Behavioral
- Control (Active Comparator): Both the control and the intervention groups will be guided in implementing structured social interaction.In the control group, the structured interaction will consist of predominantly social activities such as the caregiver reading or singing to the baby. The duration of the structured activities for both groups will be the same.
  Interventions: Other: Exercise/Social Behavioral

INTERVENTIONS:
Other: Exercise/Social Behavioral — Both the control and the intervention groups will be guided in implementing structured social interaction. In the intervention group, the structured interaction will incorporate augmented physical activities, while in the control group, the structured interaction will consist of predominantly social activities such as the caregiver reading or singing to the baby. The duration of the structured activities for both groups will be the same.

SUMMARY:
This research consists of a novel intervention designed to increase physical activity of premature babies in their first year of life. The potential beneficial impact of augmented physical activity on:

1. Body composition
2. Associated biochemical and cellular mechanisms of growth and inflammation
3. Quality of maternal care will be measured

DETAILED DESCRIPTION:
Premature birth is recognized as the single most important health problem in maternal child health in the US. Paradoxically, both failure to thrive and obesity are now known to be associated with prematurity, as are osteopenia (a condition where bone mineral density is lower than normal) and increased risk of fracture, and increased risk of cardiovascular disease later in life. We lack cohesive approaches to mitigate these profound threats to health. Despite promising new research demonstrating that physical activity can stimulate the growth of muscle and bone even during intrauterine life (perhaps through metabolic programming), there have been very few attempts to implement and study physical activity interventions in the premature baby.

The challenges are substantial and include:

* measuring body composition
* assessing physical activity
* engaging caregivers as partners in the intervention
* identifying plausible and testable biological mechanisms
* designing interventions that actually increase physical activity and match the rapid pace of motor development early in life

A developmentally dynamic physical activity intervention has been designed and pilot tested-one that engages the caregiver as a partner. Using techniques and tools as far-ranging as Dual X-ray Absorbiometry (DXA), smart phones, doubly labeled water, and lightweight, wireless accelerometers developed specifically for this purpose, the working hypothesis is that the one-year intervention will augment lean body mass (primary outcome variable) and improve bone mineralization and the ratio of lean to fat tissue (secondary outcome variables). The study will gauge the impact of the physical activity intervention on the balance between circulating anabolic mediators (insulin-like growth factor-I and growth hormone binding protein) and inflammation-associated cytokines (interleukin-6, and interleukin-1 receptor antagonist), which antagonize muscle and bone growth.

We will additionally:

1. begin to explore how physical activity influences circulating endothelial progenitor cells, which are increasingly viewed as markers of vascular health very early in life
2. take advantage of this prospective, interventional study to explore potential genetic determinants of growth in babies born prematurely.
3. Finally, any study involving the premature infant and the data associated with it must be viewed in light of the critical relationship between the mother and baby.

The potential broad impact of early life interventions has been recently demonstrated by the success of the "Back-To-Sleep" campaign in mitigating sudden infant death syndrome. Should the positive effects of augmented exercise on body composition be supported, we would then anticipate widespread benefit in preventing long-term health consequences of prematurity at relatively low cost.

ELIGIBILITY:
Infant Inclusion criteria:

* Infant is a healthy, growing NICU inpatient.
* Caregiver ≥18 years of age
* Infant gestational age at birth <29weeks
* Infant gestational age at time of study recruitment >34 wks, on full feeds and nearing discharge

Infant Exclusion criteria:

* Significant lung disease of prematurity requiring supplemental oxygen or corticosteroids at discharge
* Significant intraventricular hemorrhage, grade III -IV
* Necrotizing entrocolitis
* Tracheostomy
* Bone Diseases

  * Osteogenesis Imperfecta
  * Hip or knee joint anomalies
  * Arthrogryposis
  * Fractures
* Skin disorders (e.g., Erythematus Bullosis)
* Symptomatic congestive heart disease
* Any other conditions or congenital anomalies likely to severely impact the ability of the premature baby and caregiver to participate in a demanding study

Ages: 29 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in Lean Body Mass (LBM) as assessed by Dual X-ray Absorbiometry(DXA) at age 34-40 weeks gestational age and 86-92 weeks of age | ages: 34-40 weeks gestational age and 86 - 92 weeks of age
  LBM (lean body mass) will be measured and compared at the UCI Institute for Clinical and Translational Science. Dual X-ray Absorbiometry (DXA) scan to measure lean mass will be done using a whole body fan-beam scanner (Hologic QDR Discovery-A Hologic Inc., Bedford MA)at age 34-40 weeks gestational age and again at 86-92 weeks of age

SECONDARY OUTCOMES:
Blood sample | ages: 34-40 weeks gestational age and 86 - 92 weeks of age
  Blood sample (IGF-I)insulin-like growth factor-I , (GHBP)growth hormone binding protein, (IL-1ra)interleukin-1 receptor antagonist,(IL-6)interleukin-6, (EPCs)Epithelial Progenitor Cells. Inflammatory/Stress and growth factors will be measured from infant blood. A blood sample will be obtained from the NICU before discharge. A second blood sample will be obtained (venous) from the infant at 1 year.The Enzyme-linked immunosorbent assay (ELISAs) for IGF-I, IL-6, GHBP, and IL-1ra are available and routinely performed in our laboratory.
Energy Expenditure 1 Accelerometer three time points in the study | ages: 34-40 weeks gestational age, 52-68 weeks and 86 - 92 weeks of age
  Accelerometers provide robust, high fidelity logging of observed limb acceleration. The devices are worn in a canonical and identical orientation relative to the anatomy of each infant. Sleep/wake cycles of the babies will be synchronized to assure that comparable activity.
Energy expenditure 2 Total Energy Expenditure as assessed by Doubly Labeled Water | age: 86-92 weeks
  A study a subset of 100 of our enrollees will have total energy expenditure assessed by DLW. DLW measurements in children will be sent to our subcontract William Wong at Baylor University
Diet Assessments | ages: 34-40 weeks gestational age, 52-68 weeks and 86 - 92 weeks of age
  Parents will be called at two random days during the week of the assessment, thereby making sure that the recall interviews capture 1 weekday and 1 weekend day. Information on infant nutrition will also be obtained by three 24-h dietary recall interviews with the primary caregiver. Each interview will take approximately 20-30 minutes.
Quality of Caregiver-Child Interaction | ages: 34-40 weeks gestational age and 86 to 92 weeks of age
  A standardized laboratory protocol developed for the National Institute of Child Health and Human Development (NICHD) Study of Early Child Care and Youth Development and used currently by our group of researchers will be administered to determine quality of maternal infant interaction. For this protocol, observations are made during semi-structured play.
TIMP/AIMS | ages: 34-40 weeks gestational age and 86 to 92 weeks of age
  TIMP(Test of Infant Motor Performance)/AIMS(Alberta Infant Motor Scale) The AIMS (Alberta Infant Motor Scale) is a reliable norm-referenced observational motor assessment. The AIMS measures qualitative aspects of movement and it is sensitive to changes in infant's motor performance. We also plan a test of motor development (TIMP, Test of Infant Motor Performance) that was developed specifically for newborns, overlaps well with the AIMS, and can be used to guide our exercise intervention in the first months of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dan M. Cooper, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Douglas Hospital, Orange, California, United States